CLINICAL TRIAL: NCT01612091
Title: The Monitoring Messenger: Mobile Patient Monitoring for the Pediatric Intensive Care Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced with updated protocol as H16-02361
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Ansermino, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H12-01270
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Medical Device; User-Computer Interface; Critical Care; Physiologic Monitoring
Keywords: Expert System; Intensive Care; Telemedicine; Equipment Design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring Messenger (Experimental)
  Interventions: Device: Monitoring Messenger
- Control (Active Comparator): Traditional tools (monitors, paper records)
  Interventions: Device: Traditional tools

INTERVENTIONS:
Device: Monitoring Messenger — Monitoring Messenger prototype device
  Arms: Monitoring Messenger
Device: Traditional tools — Paper based records, screenshots of monitors and therapy devices
  Arms: Control

SUMMARY:
The Mobile Messenger is a unified, portable and intelligent device that integrates information from multiple patient monitors, mechanical ventilators, infusion pumps and clinical information systems on a mobile platform. It will allow nurses, respiratory therapists and physicians to continuously monitor and coordinate care of critically ill patients. This study will use a participatory design process to guide the design of an integrated mobile device. Next, we will evaluate the proposed device in a simulated ICU setting.

DETAILED DESCRIPTION:
There are a limited number of nurses, respiratory therapists and physicians in an ICU at a given time. To make decisions and plan therapies, these clinicians need to observe, assimilate and interpret a vast array of information originating from various devices located on the bedsides of multiple patients. Several shortcomings in existing technology limit their abilities: a) the fixed location of monitoring devices at the bedside; b) information overload from a multitude of devices, each with its own display; c) the lack of integration and interaction between these devices; d) the use of visually cumbersome displays, which were historically created for monitoring during anesthesia but never optimized for users in the ICU; and e) lack of context specific information (such as historical trends) to support patient data interpretation and clinical decision making.

This project proposes to address these challenges in ICU monitoring by developing a unified, portable, and intelligent device: the Monitoring Messenger. By integrating information from multiple monitoring devices, mechanical ventilators, infusion pumps and clinical information systems on a mobile device (tablet PC or smart phone); the Monitoring Messenger will allow nurses, respiratory therapists and physicians on or off-site, to continuously monitor critically ill patients, thereby increasing patient safety.

The proposed experiment will have two parts: Part I - Participatory design and Part II - Simulation Experiment.

In Part I - Participatory Design. Participatory design an inter-professional team of nurses, physicians, designers, engineers, and human factors experts will follow a user-centered design process to obtain the system requirements, and obtain feedback during the rapid prototyping phase of prototype development. While we expect the resulting prototype to be easy to use, support decision making, improve awareness of the patient's condition by health care providers and reduce mental workload, this methodology is not hypothesis driven.

Part II - Simulation Experiment. In simulated ICU scenarios, the critical care physicians, nurses, and respiratory therapists will prioritize the care of critically ill patients. We expect them to do so more accurately with the use of Monitoring Messenger than with their regular tool (monitors, paper records etc). A potential outcome would be a decrease in mental workload as well as an increase in situational awareness.

ELIGIBILITY:
Inclusion Criteria:

* Staff pediatric critical care physicians, pediatric critical care fellow physicians, registered pediatric nurses and respiratory therapists will be eligible to participate in this study
* Subjects willing to provide informed consent

Exclusion Criteria:

* Inability/failure to provide informed consent.
* Nursing students and resident physicians are not eligible
* For Part II - Simulation Experiment only: Failure to complete the post-training quiz more than twice.
* Evaluation will be immediately discontinued at request of subject at any point during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of priority assignment in triaging task | Up to 1 hour
  Accuracy will be measured by matching of the participants triage priority ranking with the previously defined expert ranking.

SECONDARY OUTCOMES:
Requirements for design of the mobile device | Up to 2 hours
  Information requirements for tasks, task frequencies, perceived challenges and potential suggestions to improve their current work environment using a mobile monitoring and messaging device

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ansermino, MBBCh, FRCPC, Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada